CLINICAL TRIAL: NCT01142024
Title: Polymorphism of Oxidative Stress Relative Genes in Contrast Medium Induced Nephropathy:Implications in the Pathogenesis and the Effect of Antioxidant prevention-a Prospective,Randomized,Controlled Study
Brief Title: Polymorphism of Oxidative Stress Genes in the Pathogenesis and Antioxidant Prevention of Contrast Induced Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Department of cardiology and nephrology,Huashan Hospital, HMShi,FDing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY2009-296
Record Dates: First submitted 2010-06-08; First posted 2010-06-11 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2009-12

CONDITIONS: Nephropathy; Oxidative Stress
Keywords: contrast medium induced nephropathy; polymorphism of oxidative stress genes; antioxidant prevention
MeSH Terms: conditions — Kidney Diseases | interventions — Glutathione; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- saline (Placebo Comparator): saline hydration
  Interventions: Drug: saline
- Glutathione (Experimental)
  Interventions: Drug: Glutathione

INTERVENTIONS:
Drug: Glutathione — NS 500ml + Glutathione 1.8g intravenously guttae 1-1.5ml/kg per hour,30 minutes before and during coronary angiography
  Other Names: brand name:Gluthion; serial numbers:H20040005; manufacturer:Pharminvest SPA
  Arms: Glutathione
Drug: saline — NS 500ml intravenously guttae 1-1.5ml/kg per hour,30 minutes before and during coronary angiography
  Arms: saline

SUMMARY:
With the wide use of contrast agents in clinical diagnosis and treatment, contrast induced nephropathy(CIN) accounts for 1/3 of hospital acquired acute renal failure.The mortality rate of patients with CIN is up to 35%,and about 30% patients with permanent renal dysfunction.Prevention and treatment of this iatrogenic complication and reducing morbidity has become an urgent task to every medical worker.

Now the pathogenesis of CIN is not clear,while the toxicity of renal tubular epithelial cell and the hypoxia of renal medullary is likely to be the main mechanism of CIN.Iodine contrast agent concentrate in the tubular and collecting duct and directly damage cells,leading to tubular cell death;also induce the release of renal vasoconstrictors,such as adenosine, endothelin, causing acute vasoconstriction.Furthermore,oxidative stress and the inflammatory response induced by ischemia may worsen kidney function.

Thus a large number of studies focus on oxidative stress in the pathogenesis of CIN.Recently,some studies have shown that oxidative stress proteins play an important role in acute renal injury(AKI),and have reported that these proteins of different genotypes related to the incidence and prognosis of AKI.

Therefore,the investigators speculate whether some patients have genetic potential of increased oxidative stress,and are more prone to contrast induced nephropathy? At present,there are a great number of researches about preventive measures of CIN.The firstly and widely used therapy is hydration.But it just dilutes iodine contrast medium in renal tubular and collecting duct,increases urine output to prevent the formation of tubular crystals.According to the pathogenesis of CIN,oxidative stress plays an important role in CIN,thereby several antioxidants,such as N-acetyl cysteine or Glutathione are also under study.But results are inconsistent.

As a result,the investigators designed this study to evaluate the oxidative stress in cardiovascular population on the impact of contrast medium nephropathy,and the relationship in antioxidant enzymes with genetic polymorphisms,to find clinical indicators predicting renal dysfunction and guiding individual treatment to prevent its occurrence.

DETAILED DESCRIPTION:
With the wide use of contrast agents in clinical diagnosis and treatment, contrast induced nephropathy(CIN) accounts for 1/3 of hospital acquired acute renal failure,leading to prolonged hospital stay and increased medical costs.The mortality rate of patients with CIN is up to 35%,and about 30% patients with permanent renal dysfunction.Prevention and treatment of this iatrogenic complication and reducing morbidity has become an urgent task to every medical worker.

Now the pathogenesis of CIN is not clear,while the toxicity of renal tubular epithelial cell and the hypoxia of renal medullary is likely to be the main mechanism of CIN.Iodine contrast agent concentrate in the tubular and collecting duct and directly damage cells,leading to tubular cell death;also induce the release of renal vasoconstrictors,such as adenosine, endothelin, causing acute vasoconstriction.Furthermore,oxidative stress and the inflammatory response induced by ischemia may worsen kidney function.

Thus a large number of studies focus on oxidative stress in the pathogenesis of CIN.Recently,some studies have shown that oxidative stress proteins,such as the NADPH oxidase p22 phox subunits,promote oxidase,antioxidant enzymes catalase,hypoxia inducible factor-1(HIF-1),play an important role in acute renal injury(AKI),and have reported that these proteins of different genotypes related to the incidence and prognosis of AKI,such as the NADPH oxidase subunit p22 phox (position point of +242 T replaced C).

Therefore,the investigators speculate whether some patients have genetic potential of increased oxidative stress,and are more prone to contrast induced nephropathy? At present,there are a great number of researches about preventive measures of CIN.The firstly and widely used therapy is hydration.But it just dilutes iodine contrast medium in renal tubular and collecting duct,increases urine output to prevent the formation of tubular crystals.According to the pathogenesis of CIN,oxidative stress plays an important role in CIN,thereby several antioxidants,such as N-acetyl cysteine (NAC) or Glutathione are also under study.But results are inconsistent.

As a result,the investigators designed this prospective, randomized,controlled study to evaluate the oxidative stress in cardiovascular population on the impact of contrast medium nephropathy,and the relationship in antioxidant enzymes with genetic polymorphisms,to find clinical indicators predicting renal dysfunction and guiding individual treatment to prevent its occurrence.

Inclusion Criteria:

* receiving cardiovascular angiography; age 18 to 80 years ; signed informed consent.

Exclusion Criteria:

* serum creatinine level greater than 8 mg / dL (707 μmol / L); change in serum creatinine of 0.5 mg / dL (44.2 μmol / L) or more in the 24 hours before randomization; dialysis, multiple myeloma, pulmonary edema, uncontrolled hypertension, emergency cardiac catheterization, exposure to radiographic contrast media within the preceding 2 days, allergy to radiographic contrast media, pregnancy and breast-feeding women, acceptance of mannitol and other anti-oxidant treatment.

ELIGIBILITY:
Inclusion Criteria:

* receiving cardiovascular angiography;
* age 18 to 80 years ;
* signed informed consent.

Exclusion Criteria:

* baseline serum creatinine level > 8 mg / dL (707 μmol / L);
* an increase in serum creatinine of 0.5 mg / dL (44.2 μmol / L) or more in the 24 hours before angiography;
* dialysis;
* multiple myeloma;
* pulmonary edema;
* uncontrolled hypertension;
* emergency cardiac catheterization;
* exposure to radiographic contrast media within the preceding 2 days;
* allergy to radiographic contrast media; pregnancy and breast-feeding women; acceptance of mannitol and other anti-oxidant treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Serum creatinine | 48-72h after coronary angiography
  CIN is defined as a relative increase of the serum creatinine by 25% or as an absolute increase of 0.5mg/dl(44.2umol/l) from baseline within 48-72h after contrast exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Haiming Shi, Professor, Principal Investigator — Huashan Hospital
Locations (1):
- Department of cardiology and nephrology,Huashan Hospital, Shanghai, Shanghai Municipality, China